CLINICAL TRIAL: NCT03752398
Title: A Phase 1 Multiple-Dose Study to Evaluate the Safety and Tolerability of XmAb®23104 in Subjects With Selected Advanced Solid Tumors
Brief Title: A Study of XmAb®23104 in Subjects With Selected Advanced Solid Tumors (DUET-3)
Acronym: DUET-3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XmAb23104-01; DUET-3 (Other: Xencor, Inc.)
Record Dates: First submitted 2018-11-20; First posted 2018-11-26 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Melanoma (Excluding Uveal Melanoma); Cervical Carcinoma; Pancreatic Carcinoma; Breast Carcinoma That is Estrogen Receptor, Progesterone Receptor, and Her2 Negative; Hepatocellular Carcinoma; Urothelial Carcinoma; Squamous Cell Carcinoma of the Head and Neck; Nasopharyngeal Carcinoma; Renal Cell Carcinoma; Colorectal Carcinoma; Endometrial Carcinoma; Non-small Cell Lung Carcinoma; Small Cell Lung Cancer; Gastric or Gastroesophageal Junction Adenocarcinoma; Advanced Solid Tumors; Undifferentiated Pleomorphic Sarcoma
Keywords: DUET-3; Advanced solid tumors; Melanoma; Cervical Cancer; Pancreatic Cancer; Triple Negative Breast Cancer; Hepatocellular/Liver Cancer; Urothelial Cancer; Bladder Cancer; Renal Cell Cancer; Head and Neck Cancer; Colorectal Cancer; Endometrial Cancer; Non-small Cell Lung Cancer; Small Cell Lung Cancer; Gastric Cancer; Gastroesophageal Junction Cancer; Sarcoma
MeSH Terms: conditions — Melanoma; Uterine Cervical Neoplasms; Pancreatic Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Transitional Cell; Squamous Cell Carcinoma of Head and Neck; Nasopharyngeal Carcinoma; Carcinoma, Renal Cell; Colorectal Neoplasms; Endometrial Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Histiocytoma, Malignant Fibrous; Triple Negative Breast Neoplasms; Liver Neoplasms; Urinary Bladder Neoplasms; Head and Neck Neoplasms; Stomach Neoplasms; Sarcoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XmAb®23104 Monotherapy (Experimental): XmAb®23104 administered by IV dosing on Days 1 and 15 of each 28-day cycle x 2 cycles
  Interventions: Biological: XmAb®23104
- XmAb®23104 Combination Therapy with Ipilimumab (Experimental): XmAb®23104 administered by IV on Days 1 and 15 of each 28-day cycle x 2 cycles + Yervoy® (ipilimumab)
  Interventions: Biological: XmAb®23104; Biological: Yervoy® (ipilimumab)

INTERVENTIONS:
Biological: XmAb®23104 — Monoclonal bispecific antibody
Biological: Yervoy® (ipilimumab) — Monoclonal antibody
  Arms: XmAb®23104 Combination Therapy with Ipilimumab

SUMMARY:
This is a Phase 1, multiple dose, ascending dose escalation study to define a MTD/RD and regimen of XmAb23104, to describe safety and tolerability, to assess PK and immunogenicity, and to preliminarily assess anti-tumor activity of XmAb23104 monotherapy and combination therapy with ipilimumab in subjects with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects in Part A (dose escalation) must have a diagnosis of any of the following:

   Histologically or cytologically confirmed advanced solid tumors, including the following:
   1. Melanoma (excluding uveal melanoma)
   2. Cervical carcinoma
   3. Pancreatic carcinoma
   4. Breast carcinoma that is estrogen receptor, progesterone receptor, and Her2 negative
   5. Hepatocellular carcinoma
   6. Urothelial carcinoma
   7. Squamous cell carcinoma of the head and neck
   8. Nasopharyngeal carcinoma
   9. Renal cell carcinoma
   10. Colorectal carcinoma
   11. Endometrial carcinoma
   12. NSCLC
   13. Small cell lung cancer
   14. Gastric or gastroesophageal junction adenocarcinoma
   15. Sarcoma
2. Subjects in Part B (expansion) must have a diagnosis of any of the following:

   Histologically or cytologically confirmed advanced solid tumors of the following types:
   1. Non-squamous NSCLC
   2. Melanoma
   3. HNSCC, including NPC
   4. CRC
   5. UPS, including other select high grade STS, such as MFS
   6. ccRCC

   Prior to enrolling into Part B (expansion), subjects should have received disease-specific standard therapy as indicated for:
   1. Non-squamous NSCLC
   2. Melanoma
   3. HNSCC, including NPC
   4. CRC
   5. UPS, including other select high-grade STS such as MFS
   6. RCC, clear cell histology (ccRCC)
3. Subjects in Part C (expansion)must have a diagnosis of MSS or proficient mismatch repair CRC with the following:

   1. cancer must have progressed after treatment with standard/approved therapies or have no appropriate available therapies
   2. subjects will have life expectancy greater than 3 months
4. All subjects' cancer must have progressed after treatment with standard/approved therapies or have no appropriate available therapies.
5. Subjects must have measurable disease by RECIST 1.1.
6. All subjects must have adequate archival tumor sample (slides or archival FFPE block[s] containing tumor.
7. All subjects in Part B (dose expansion) must have a tumor lesion that can be biopsied at acceptable risk (in the judgment of the Investigator) and must agree to both a fresh biopsy during screening and a second biopsy following treatment.
8. Subjects have an ECOG performance status of 0-1.

Exclusion Criteria:

1. Currently receiving other anticancer therapies
2. Prior treatment with an investigational anti-ICOS therapy
3. Treatment with any PDL1 or PDL2-directed therapy within 4 weeks of the start of study drug
4. Treatment with nivolumab within 4 weeks of the start of study drug
5. Treatment with pembrolizumab within 24 weeks of start of study drug for Cohorts 1A - 10A
6. Treatment with any other anticancer therapy within 2 weeks of the start of study drug (ie, other immunotherapy, chemotherapy, radiation therapy, etc.)
7. A life-threatening (Grade 4) irAE related to prior immunotherapy
8. Failure to recover from any irAE from prior cancer therapy to Grade ≤ 1, except for endocrinopathies that are on stable hormone replacement doses
9. Failure to recover from any other toxicity (other than immune-related toxicity) related to previous anticancer treatment to Grade ≤ 2
10. Known active central nervous system involvement by malignant disease. Subjects with previously treated brain metastases may participate provided they are radiologically stable, ie, are without evidence of progression for at least 4 weeks by repeat imaging and are clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
11. Active known or suspected autoimmune disease
12. Receipt of an organ allograft
13. History or evidence of any other clinically unstable/uncontrolled disorder, condition, or disease (including, but not limited to, cardiopulmonary, renal, metabolic, hematologic or psychiatric) other than their primary malignancy, that in the opinion of the Investigator would pose a risk to patient safety or interfere with study evaluations, procedures, or completion
14. Treatment with antibiotics within 14 days prior to first dose of study drug
15. Receipt of a live-virus vaccine within 30 days prior to first dose of study drug (seasonal flu vaccines that do not contain live virus are permitted).
16. Treatment with ipilimumab within 4 weeks of the start of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Treatment-related adverse events as assessed by CTCAE v4.03 | 56 Days
  Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Chet Bohac, MD, MSc, Study Director — Xencor, Inc.
Locations (18):
- United States (18):
  - UC San Diego Moores Cancer Center, San Diego, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Emory University, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research - Medical City, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No